CLINICAL TRIAL: NCT07044661
Title: Effect of Bilateral vs. Unilateral Alveolar Recruitment on Gas Exchange in Lung Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2025-0522
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer Requiring Surgical Resection Under One-lung Ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uni-ARM group (Active Comparator): Unilateral ARM is performed immediately after lateral decubitus positioning of the patient, followed by lung-protective mechanical ventilation with individualized PEEP.
  Interventions: Procedure: Unilateral ARM
- Bi-ARM group (Experimental): Bilateral ARM is performed immediately after lateral decubitus positioning of the patient, followed by lung-protective mechanical ventilation with individualized PEEP.
  Interventions: Procedure: Bilateral ARM

INTERVENTIONS:
Procedure: Unilateral ARM — ARM is performed to the dependent lung only. During ARM, mechanical ventilation is set to a pressure-controlled ventilation mode with a driving pressure of 20 cmH₂O and an inspiratory-to-expiratory ratio of 1:1. The positive end-expiratory pressure (PEEP) is increased by 5 cmH₂O every five respiratory cycles, reaching a final PEEP of 20 cmH₂O and a peak airway pressure of 40 cmH₂O, which is then maintained for ten respiratory cycles.
  Arms: Uni-ARM group
Procedure: Bilateral ARM — ARM is performed to both lungs. During ARM, mechanical ventilation is set to a pressure-controlled ventilation mode with a driving pressure of 20 cmH₂O and an inspiratory-to-expiratory ratio of 1:1. The positive end-expiratory pressure (PEEP) is increased by 5 cmH₂O every five respiratory cycles, reaching a final PEEP of 20 cmH₂O and a peak airway pressure of 40 cmH₂O, which is then maintained for ten respiratory cycles.
  Arms: Bi-ARM group

SUMMARY:
"One-lung ventilation (OLV) is an essential technique during thoracic surgery but preventing atelectasis during OLV remains a key challenge in thoracic anesthesia.

Several previous randomized controlled trials have demonstrated that alveolar recruitment maneuvers (ARMs) can significantly reduce driving pressure, peak airway pressure, plateau pressure, and anatomical dead space. However, the optimal method for implementing ARMs has not yet been standardized, as the timing and target of ARM application vary among studies. Some protocols involve applying ARMs to both lungs immediately prior to the initiation of OLV (bilateral ARM), while others apply ARMs solely to the non-operative lung after OLV has begun (unilateral ARM). Bilateral ARM may provide prolonged improvement in gas exchange but carry the risk of insufficient collapse of the operative lung. Conversely, unilateral ARM may facilitate better collapse of the operative lung compared to bilateral ARMs, though potentially at the expense of gas exchange. To date, no study has directly compared these two approaches. This study aims to compare and evaluate the effects of bilateral versus unilateral ARM performed immediately prior to thoracic incision on intraoperative gas exchange and the incidence of intraoperative and postoperative complications."

ELIGIBILITY:
Inclusion Criteria:

* -Adult patients aged 20 to 80 years scheduled for thoracoscopic lung resection.
* American Society of Anesthesiologists (ASA) physical status classification of I to III.

Exclusion Criteria:

* Anticipated duration of one-lung ventilation (OLV) less than 1 hour.
* Diagnosis of heart failure.
* History of pneumothorax or radiologic evidence of pulmonary blebs or bullae prior to surgery.
* Patients receiving supplemental oxygen therapy or mechanical ventilation prior to surgery.

Dropout Criteria

* Actual duration of OLV less than 1 hour.
* Surgery is canceled or converted to an open thoracotomy or another surgical approach.
* Inability to maintain peripheral oxygen saturation ≥90% despite adjustments in inspired oxygen fraction.
* Inability to maintain ventilator settings due to extensive pulmonary adhesions.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
PaO₂/FiO₂ at 60 minutes after ARM | PaCO₂ is assessed by arterial blood gas analysis at 60 minutes after ARM.
  We analyze whether different methods of ARM result in significant differences in the PaO₂/FiO₂ ratio measured at 60 minutes after the initiation of one-lung ventilation (OLV60).

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Severance hospital, Seoul

IPD SHARING:
Plan to Share IPD: No